CLINICAL TRIAL: NCT06658574
Title: Comparative Efficacy of Two Different Oral Dosage Forms of Acetaminophen for Post-operative Analgesia in Bariatric Surgery Patients
Brief Title: Oral Acetaminophen for Post-Op Pain Management in Bariatric Surgery Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Robert Wood Johnson Medical School (Other)
Responsible Party: Principal Investigator, Daniel T. Abazia, PharmD, Clinical Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro2023002382
Record Dates: First submitted 2024-10-16; First posted 2024-10-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Analgesia; Bariatric Surgery; Bariatric Surgery (Gastric Bypass); Bariatric Surgery Patients; Perioperative Analgesia
Keywords: Acetaminophen; Bariatric; Analgesia; Perioperative; Post Operative
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Oral acetaminophen - Tablet (Experimental): Acetaminophen 650 mg tablet by mouth
  Interventions: Drug: Acetaminophen
- Oral acetaminophen - Liquid (Experimental): Acetaminophen 650 mg liquid by mouth
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Arm 1: Once cleared for oral intake - acetaminophen tablets 650 mg PO every 6 hours PRN - mild pain (1 - 3) to a maximum of 4 grams daily for 3 days' dispensed as unit-dose tablets Arm 2: Once cleared for oral intake - acetaminophen liquid (160 mg/5 mL) 650 mg PO every 6 hours PRN - mild pain (1 - 3) to a maximum of 4 grams daily for 3 days; 650 mg = 20.3 mL, dispensed as a unit-dose cup

SUMMARY:
Adult patients with morbid obesity who have had Roux-en-Y gastric bypass (RYGB) or laparoscopic sleeve gastrectomy (LSG) surgery have impaired drug metabolism. There is a paucity of information available on how these patients metabolize acetaminophen post operatively and if drug preparation has any effect on achieving adequate pain control. The surgery may alter the stomach pH, reduce surface area of the stomach, affect transit time, and alter anatomic and physiologic standard absorption of medications. Due to these anatomic and physiologic changes, we seek to understand the potential effects of liquid versus pill formulations of acetaminophen on pain control in this patient population. The purpose of this study is to assess for subjective and objective measures of optimized pain control between formulations of acetaminophen including oral pills and oral liquid.

DETAILED DESCRIPTION:
There is limited information on pharmacokinetics among morbidly obese patients and even less among patients who have undergone metabolic and bariatric surgery (MBS). However, it is known that these patients have altered metabolism due to anatomic and physiologic changes related to body habitus, that are further complicated post MBS. The quadruple aim consists of population health, reduces costs, improved healthcare worker experience and improved patient experience. To provide a comprehensive healthcare approach for this patient population, improved pain management through the utilization of lower cost formulations of acetaminophen can result in improved patient experience through enhanced pain management, avoidance of unnecessary ED visits and/or hospital readmissions. Healthcare worker experience may be improved through less provider and nurse burden from under managed pain, and improved patient outcomes resulting in greater job satisfaction. In 2021, the annual drug overdose death rate in New Jersey is 32.4 per 100,000.3 It is essential that alternatives to opioid medications provide adequate pain control if we are to address this public health crisis.

No previous research was identified that evaluates the effectiveness of tablet vs liquid oral acetaminophen despite some evidence of alterations in absorption of tablets among post RYGB or LSG patients. In a small study among severely obese adolescent females, results demonstrated the participants required more than double the amount of IV acetaminophen to achieve equal serum concentrations. Additionally, a small study demonstrated that to achieve near-equivalent pain control post-operatively of colorectal surgery, IV acetaminophen was more effective when administered. Additional studies have demonstrated increased clearance of drugs metabolized by CYP1A2 and CYP2D6 pathways. These pathways are specifically involved in acetaminophen metabolism. The main pathway for acetaminophen metabolism is glucuronidation. Obesity has been associated with increase glucuronide clearance, therefore leaving less acetaminophen available for metabolism by CYP2E1. Furthermore, the anatomic and physiologic changes post-operatively, including a decrease gastrointestinal surface area and length contribute to alternations in drug bioavailability. This evidence leads to the hypothesis that higher dosing of oral acetaminophen is required to achieve adequate pain control when compared to non-obese patients. Based upon previous literature and current understanding of post-operative anatomic and physiologic alterations, there is a lack of evidence to support the preferred formulation of oral acetaminophen in this patient population.

Objective:

To evaluate the therapeutic effects on pain control of acetaminophen pills vs. acetaminophen liquid on post-operative pain control in patients status post RYGB or LSG.

Hypotheses/Research Question(s):

H0: There will be no difference in pain control between the liquid and pill formulations of acetaminophen among patients status post RYGB or LSG.

H1: The investigators hypothesize that based on post-operative changes, the liquid formulation of acetaminophen will result in improved pain control among patients status post RYGB or LSG.

Research Procedures:

Prior to initiation of the study, pharmacy, nursing, and medical leadership will be informed of the stratification of acetaminophen formulations based upon surgery day.

Patients will be stratified to two arms of the study utilizing the National Cancer Institute's Clinical Trial Randomization Tool. Trial parameters using the asymptotic maximal randomization method, ratio of 1:1, and a participant count of 150 were inputted to create a randomization file. Presently, all patients receive acetaminophen as part of their multi-modal post-operative pain management. The clinical coordinator of the bariatric program on this study will recruit patients during the pre-operative admission process. Consent will occur at the bedside in same day surgery. The clinical coordinator for the bariatric program who is a study team member will be responsible for obtaining patient consent into the study. It is anticipated the consent discussion will be less than 15 minutes per patient. There is no waiting period expected.

It is anticipated that equal number of patients in both arms of the study will be obtained.

Data Points:

Variable will include length of stay (LOS), morphine equivalents, documented pain level, heart rate after cleared from anesthesia, blood pressure after cleared from anesthesia, ED visits within 7 days from discharge, hospital readmissions within 7 days, out of bed/ambulation, time to PO acetaminophen. Demographic data including age, sex, race, weight, height, BMI, co-morbidities.

Study Duration:

The enrollment period is anticipated to be three months. Total study duration, including data analysis and manuscript writing are anticipated to take two years.

Endpoints:

Participants may be removed from the study if experiencing inadequate pain control or experiencing elevated glucose levels to ensure pain control and glucose are medically managed as required. Participants will be removed from the study if they experience any allergic reactions to any formulation of acetaminophen to ensure patient safety.

Primary outcomes include pain control. Secondary outcomes include LOS and morphine equivalents.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years old or greater who meet patient selection criteria for either primary Roux-en-Y gastric bypass or primary laparoscopic sleeve gastrectomy.

Exclusion Criteria:

* Patients with a known hypersensitivity or history of intolerance to acetaminophen or any inactive ingredients in either formulation. Patients uncomfortable with or unable to take pills.
* Surgical: Duodenal Switch (DS) surgeries, Adjustable Gastric Banding (AGB), surgical revisions, and surgical conversions.
* Medical: patients with documented history of chronic and/or current pain syndrome, as evidenced by documentation of ICD-10 code G89.4, patients with documented ICD-10 code F11.90, indication unspecified, uncomplicated opioid use.
* Patients of vulnerable populations, as outlined by federal guidelines as children, prisoners, pregnant women, and mentally disabled persons will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pain control | From date of consent until the date of hospital discharge, assessed up to 3 months.
  Numeric Rain Scale (The scale has a fixed range with 0 representing "no pain" and the upper limit of 10 representing "worst pain possible")

SECONDARY OUTCOMES:
Length of stay (LOS) | From date of consent until the date of hospital discharge, assessed up to 3 months
  Participants' length of hospital stay in days.
Milligrams Morphine Equivalents (MME) | From date of consent until the date of hospital discharge, assessed up to 3 months
  Values that represent the potency of an opioid dose relative to morphine.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Abazia, PharmD, BCPS, CPPS, Principal Investigator — Rutgers University - Ernest Mario School of Pharmacy
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No